CLINICAL TRIAL: NCT02907632
Title: Use of Metoclopramide for the Prevention of Gastroesophageal Reflux in Premature Infants Followed in an Outpatient Kangaroo Mother Care Clinic Before 40 Weeks of Gestational Age: A Randomized Controlled Trial
Brief Title: Methoclopramide for Gastroesophageal Reflux in Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nathalie Charpak (Other)
Collaborators: Hospital Universitario San Ignacio (Other); Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor-Investigator, Nathalie Charpak, Doctor, Kangaroo Foundation
Organization: Kangaroo Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015/71
Record Dates: First submitted 2016-09-13; First posted 2016-09-20 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Gastroesophageal Reflux
Keywords: Metoclopramide; Pro kinetic; Gastroesophageal Reflux; Premature Infant; Low Birth Weight; Kangaroo Mother Care Method
MeSH Terms: conditions — Gastroesophageal Reflux; Premature Birth | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoclopramide (Experimental): Blind and randomized allocation to the experimental treatment: Metoclopramide
  Interventions: Drug: Metoclopramide
- Placebo (Placebo Comparator): Blind and randomized allocation to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide — Metoclopramide Solution 4 mg / ml; 30 ml canister (1 drop equals 0.2 mg). Dose: 0.2 mg / kg / dose (1 drop per kg) every 8 hours orally 15 minutes before lactation.
  Duration: Until the child completes 40 weeks of post menstrual age.
  Other Names: Plasil
  Arms: Metoclopramide
Drug: Placebo — Oral solution: 1 drop per kg of placebo 15 minutes before lactation with identical presentation appearance, taste and color than Metoclopramide. Duration: Until the child completes 40 weeks of post menstrual age.
  Arms: Placebo

SUMMARY:
Gastroesophageal Reflux (GER) is a condition that affects the majority of premature infants that are followed at the Kangaroo Mother Care Program (ambulatory program for preterm infants discharged with their mothers in continuous skin to skin contact and strict outpatient follow up). For over 20 years, the use of Metoclopramide has been systematic among all preterm infants according to the protocols of the Kangaroo Mother Care (KMC) Program . The aim of this clinical trial is to evaluate the effectiveness and security of metoclopramide to lessen the symptoms of GRE in premature infants that are followed and treated in the Ambulatory KMC Program before 40 weeks of gestational age. Design: Randomized, double blind trial, controlled with placebo. Eligible Population: Premature infants that are followed and treated in the Ambulatory Kangaroo Mother Care Program at Hospital Universitario San Ignacio before 40 weeks of gestational age, which systematically receive: metoclopramide 0.2 mg per kg, every 8 hours, 15 minutes before every feeding up to 40 weeks of gestational age, between January 01 2017 and December 31 2017.Outcomes: Incidence of regurgitation episodes reported by the parents of the infants, episodes of apnea, bronchoaspiration, postprandial irritability, the infant rejects feeding, alteration in the postprandial posture and the frequency and severity of adverse effects associated with the use of Metoclopramide such as extrapyramidal symptoms and sedation. In the case of continuous variables, the mean and median will be compared according to the distribution and for nominal variables, a chi squared test or fisher test will be carried out.

Duration: 12 months. Ethical Aspects: Experiment with minimum mayor risk. Informed consent will be requested to parents. An independent committee from the work group will be in charge of carrying out the follow-up of the safety and progression of the study. A methodological expert, a thematic expert, a statistician and an expert in bioethics will constitute the committee.

Financial Disclosure: The study will be funded through the Kangaroo Foundation with the collaboration of the " Hospital Universitario San Ignacio", Bogotá, Colombia.

DETAILED DESCRIPTION:
Justification: Gastroesophageal Reflux (GER) is a condition that affects the majority of premature infants that are followed at the Kangaroo Mother Care Program. The incidence of GRE in premature infants can oscillate between 22 and 85% depending on the criteria used to diagnose GER, which can vary among healthcare professionals.

For over 20 years, the use of metoclopramide has been systematic among all preterm infants according to the protocols of the Kangaroo Mother Care (KMC) Program. These protocols were established according to the recommendations emitted by the Cochrane Collaboration in 2006, nevertheless according to new studies published in the last years, the controversial evidence referring the use of metoclopramide given the eventual possibility of adverse effects and the lack of evidence in premature infants, it is necessary to evaluate whether it is pertinent to continue the use of metoclopramide in premature infants and the risk of adverse effects.

Objective: To evaluate the effectiveness and security of metoclopramide to lessen the symptoms of GRE in premature infants that are followed and treated in the Ambulatory KMC Program before 40 weeks of gestational age.

Design: Randomized, double blind trial, controlled with placebo. Eligible Population: Premature infants that are followed and treated in the Ambulatory KMC Program at Hospital Universitario San Ignacio before 40 weeks of gestational age, which systematically receive: metoclopramide 0.2 mg per kg, every 8 hours, 15 minutes before every feeding up to 40 weeks of gestational age, between April 1 2017 and January 31 2019. Intervention: Blind and randomized allocation to the experimental treatment (metoclopramide 0.2 mg per kg, every 8 hours, 15 minutes before every feeding up to 40 weeks of gestational age) or placebo.

Outcomes: Incidence of regurgitation episodes reported by the parents of the infants, episodes of apnea, bronchoaspiration, postprandial irritability, the infant rejects feeding, alteration in the postprandial posture and the frequency and severity of adverse effects associated with the use of metoclopramide such as extrapyramidal symptoms and sedation. In the case of continuous variables, the mean and median will be compared according to the distribution and for nominal variables, a chi squared test or fisher test will be carried out.Intervention: Blind and randomized allocation to the experimental treatment (metoclopramide 0.2 mg per kg, every 8 hours, 15 minutes before every feeding up to 40 weeks of gestational age) or placebo.

Expected Results: Reliable information regarding the use of metoclopramide in premature infants for the prevention of regurgitation episodes associated to apnea, cyanosis, irritability, rejection of feeding efforts, bronchoaspiration and poor weight gain as well as adverse effects.

Duration: 12 months. Ethical Aspects: Experiment with minimum mayor risk. Informed consent will be requested to parents. An independent committee from the work group will be in charge of carrying out the follow-up of the safety and progression of the study. A methodological expert, a thematic expert, a statistician and an expert in bioethics will constitute the committee.

Financial Disclosure: The study will be funded through the Kangaroo Foundation with the collaboration of the " Hospital Universitario San Ignacio", Bogota, Colombia.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants followed at ambulatory Kangaroo Mother Care Program(KMCP) in Hospital San Ignacio, Bogotá, Colombia.

Exclusion Criteria:

Hipoxic- Ischemic Encephalopathy. Periventricular Leukomalacia (PVL). Intraventricular hemorrhage grade 3 or 4. Severe dystonia Seizures. Liver failure. Renal insufficiency. Previous adverse events with the use of Metoclopramide. Parents don´t agree participation.

Ages: 1 Day to 100 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 490 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of regurgitation episodes | Until 40 weeks Post Menstrual Age
  Reported by the parents of the infants in a diary.

SECONDARY OUTCOMES:
Episodes of apnea | Until 40 weeks Post Menstrual Age
  Reported in clinical history
Bronchoaspiration | Until 40 weeks Post Menstrual Age
  Reported in clinical history
Postprandial irritability | Until 40 weeks Post Menstrual Age
  Reported by the parents of the infants in a diary
The infant rejects feeding | Until 40 weeks Post Menstrual Age
  Reported by the parents of the infants in a diary
Alteration in the postprandial posture | Until 40 weeks Post Menstrual Age
  Reported by the parents of the infants in a diary

OTHER OUTCOMES:
extrapyramidal symptoms | Until 40 weeks Post Menstrual Age
  Reported in clinical history

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Charpak, Dr., Study Director — Kangaroo Foundation Director
Locations (1):
- Nathalie Charpak, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hibbs AM, Lorch SA. Metoclopramide for the treatment of gastroesophageal reflux disease in infants: a systematic review. Pediatrics. 2006 Aug;118(2):746-52. doi: 10.1542/peds.2005-2664. PMID 16882832
- [Result] Tighe MP, Afzal NA, Bevan A, Beattie RM. Current pharmacological management of gastro-esophageal reflux in children: an evidence-based systematic review. Paediatr Drugs. 2009;11(3):185-202. doi: 10.2165/00148581-200911030-00004. PMID 19445547
- [Derived] Montealegre-Pomar ADP, Charpak N. Randomized Clinical Trial of Metoclopramide as Prophylaxis of Gastroesophageal Reflux Disease in Preterm Infants. Paediatr Drugs. 2021 Nov;23(6):591-599. doi: 10.1007/s40272-021-00475-x. Epub 2021 Oct 25. PMID 34693501